CLINICAL TRIAL: NCT01015690
Title: Incidence of Early Pregnancy Loss in Patients With Unexplained Infertility Measured by hCG Rise in Urine
Brief Title: Incidence of Early Pregnancy Loss in Patients With Unexplained Infertility
Acronym: UNEXPLAINED
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: NS Macklon, Prof, PhD, UMCUtrecht
Other Study IDs: UNEXPLAINED
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Infertility
Keywords: unexplained infertility; hCG; early pregnancy loss
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- unexplained infertility: patients with unexplained infertility
- healthy controls: women who wish to conceive, no more tha 3 previous cycles, age above 18
- references: lesbian women with a regular cycle without use of anticonception and not at risk of becoming pregnant

SUMMARY:
Unexplained fertility could be partly caused by a higher incidence of early pregnancy loss in this group. 65 women with unexplained infertility and 65 healthy controls will collect daily urine samples form the luteal phase. hCG and creatinine levels are measured in order to detect pregnancies and early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility

Exclusion Criteria:

* IVF treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with unexplained infertility and healthy controls have collected urine samples in the luteal phase of the menstrual cycle for detection of hCG rise and pregnancy
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
incidence of early pregnancy loss | 3 mentrual cycles

SECONDARY OUTCOMES:
incidence of pregnancies | 3 menstual cycles

CONTACTS AND LOCATIONS:
Overall Officials: NS Macklon, Prof, Principal Investigator — UMC Utrecht
Locations (1):
- UMCUtrecht, Utrecht, Utrecht, Netherlands